CLINICAL TRIAL: NCT00478907
Title: phase2 Study of Prevention of Complications of Strabismus Surgery
Brief Title: Prevention of Complications of Eye Surgery
Acronym: ocr
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 82390
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2007-05-25 (Estimated); Status verified 2007-05

CONDITIONS: Strabismus
Keywords: oculocardiac reflex; strabismus surgery;
MeSH Terms: conditions — Strabismus | interventions — Ketamine; Propofol; Thiopental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: KETAMINE, PROPOFOL, THIOPENTAL

SUMMARY:
This study was designed to investigate pre-operatively measured parameters of various anaesthetic regimes, iris color, sex, age, surgical time, severity of Marcus-Gunn Pupil (MGP), type of mechanical stimulation of eye, and number of extraocular muscle (EOM) under tension as predictors of significant OCR in pediatric strabismus surgery.

DETAILED DESCRIPTION:
Objectives: Despite various proposed maneuver, successfully predicting an oculocardiac reflex (OCR) is difficult to achieve. This study was designed to investigate pre-operatively measured parameters of various anaesthetic regimes, iris color, sex, age, surgical time, severity of Marcus-Gunn Pupil (MGP), type of mechanical stimulation of eye, and number of extraocular muscle (EOM) under tension as predictors of significant OCR in pediatric strabismus surgery.

Methods: Three hundred patients were randomized to one of three anesthetic regimes: group P: propofol (2 mg/kg), alfentanil 0.02 mg/kg, and atracurium 0.5 mg/kg at induction; group K: ketamine (2mg/kg), alfentanil 0.02 mg/kg, and atracurium 0.5 mg/kg at induction; group T: thiopental (5mg/kg), alfentanil 0.02 mg/kg, and atracurium 0.5 mg/kg at induction. OCR was defined as a 10% change in heart rate induced by traction.

Results: Incidence of OCR was significantly lower in patients in group k compared with patients in group T or P. Chi-square test results showed that the occurrence of OCR was significantly associated with difference of iris color (P=0.01). The occurrence of the OCR did not correlate with sex, age, duration of surgery, iris color, severity of MGP, number of EOM under tension, and type of mechanical stimulation of eye. Type of mechanical stimulation of eye or number of EOM under tension increased risk of developing OCR by 0.81 (95% CI, 0.66-0.98) and 1.29 (95% CI; 1.12-1.63) respectively.

Conclusions: Induction of anesthesia with ketamine is associated with least hemodynamic changes induced by OCR during strabismus surgery. The prediction of oculocardiac reflex propensity remains elusive.

ELIGIBILITY:
Inclusion Criteria:

* 300 ASA physical status I or II patients, aged 2-18 years, who candidate for elective strabismus surgery

Exclusion Criteria:

* trauma to eye, ASA III or IV, who had contraindication for using thiopental, ketamine, or propofol, had cardiovascular diseases or had taken cardiovascular drugs

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 300 (Actual)
Dates: Start 2004-03; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
incidence of OCR | TWO YEARS

SECONDARY OUTCOMES:
TYPE OF DRUG PREVENTING OCR | 2 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: mohammad safavi, phd, Study Chair — isfahan committee of research; hasan soltani, phd, Principal Investigator — feiz hospital
Locations (1):
- Feiz Hospital, Tīrān, Isfahan, Iran

REFERENCES:
- [Background] Apivor D, Ravi PK. Ketamine and the oculocardiac reflex. Dysrhythmia in pediatric strabismus surgery: the role of intravenous atropine. Anaesthesia. 1976 Jan-Feb;31(1):18-22. doi: 10.1111/j.1365-2044.1976.tb11740.x. PMID 1259120
- See also: oculocardiac reflex ketamine — http://www.ncbi.nlm.nih.gov/entrez/query.fcgi?cmd=Search&db=pubmed&term=oculocardiac+reflex+ketamine&tool=fuzzy&ot=oculocardac+reflex+ketamine